CLINICAL TRIAL: NCT06395753
Title: A Phase 2, Randomized, Open-Label, Dose-Finding Study of Debio 4228, an Extended-Release Formulation of Gonadotropin-Releasing Hormone Antagonist in Participants With Advanced Prostate Cancer
Brief Title: A Dose Finding Study of Debio 4228 in Participants With Advanced Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Debio 4228-201; U1111-1298-8943 (Other: WHO Unique Trial Identifier); 2024-511038-11 (Other: EU CT Number)
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: Debio 4228 Dose Level 1 (Experimental): Participants will receive a single intramuscular (IM) administration of dose level 1 Debio 4228 on Day 1. Enrolment for cohort 1 was discontinued as per protocol amendment v5.0
  Interventions: Drug: Debio 4228
- Cohort 2: Debio 4228 Dose Level 2 (Experimental): Participants will receive a single IM administration of dose level 2 Debio 4228 on Day 1.
  Interventions: Drug: Debio 4228
- Cohort 3 (Experimental): If any alternative dose is deemed necessary based on preliminary data, participants may be enrolled in Cohort 3 to receive Debio 4228 loading dose IM, on Day 1 followed by a maintenance dose IM, 12 weeks after receiving the loading dose (Day 85).
  Interventions: Drug: Debio 4228

INTERVENTIONS:
Drug: Debio 4228 — Administered as IM injection.

SUMMARY:
The primary purpose of this study is to determine the pharmacokinetics (PK) and pharmacodynamics (PD) of Debio 4228.

ELIGIBILITY:
Inclusion Criteria:

1. Participant with histologically confirmed diagnosis of prostate cancer, with one of the following:

   1. Newly diagnosed androgen-sensitive locally advanced or metastatic disease; or
   2. Localized disease not suitable for local primary intervention with curative intent.
2. Participant judged by the Study Investigator to be candidate for continuous androgen deprivation therapy (ADT).
3. Baseline morning serum testosterone levels >150 ng/dL at screening visit.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
5. Life expectancy of at least 6 months.
6. Adequate bone marrow, hepatic, and renal function at the screening visit.

[Note: Other protocol and subprotocol-defined criteria apply]

Exclusion Criteria:

1. Previous ADT (neoadjuvant or adjuvant hormonal therapy) for ≥6 months duration and <6 months treatment-free interval before start of screening.
2. Participant requires combination with androgen deprivation therapy with the exception of enzalutamide.
3. History of bilateral orchiectomy, adrenalectomy, or hypophysectomy.
4. Received chemotherapy or cryotherapy within 8 weeks prior to the start of screening for the treatment of prostate cancer.
5. Abnormal cardiovascular function or diabetes.
6. Use of exogenous testosterone within 6 months before the start of screening.
7. Major surgery within 4 weeks before the start of screening.
8. Cancer disease within the last two years except for prostate cancer and some skin cancers.

[Note: Other protocol and subprotocol-defined criteria apply]

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males with advanced prostate cancer.
Enrollment: 66 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of Debio 4228 | Cohorts 1 and 2: Predose and at multiple time points post-dose up to Day 169; Cohort 3: Predose and at multiple time points post-dose up to Day 169
Area Under the Concentration-time Curve of Debio 4228 Over 12 weeks (AUC84d) | Cohorts 1 and 2: Predose and at multiple time points post-dose up to Day 84; Cohort 3: Predose and at multiple time points post-dose up to Day 169
Plasma Concentration of Debio 4228 at Week 12 (C84d) | Cohorts 1 and 2: Post-dose on Day 84; Cohort 3: Post-dose on Days 84 and 168
Serum Concentration of Testosterone | Cohorts 1 and 2: Predose and at multiple time points post-dose from Days 1 to 85; Cohort 3: Predose and at multiple time points post-dose from Days 1 to 169

SECONDARY OUTCOMES:
Number of Participants who Achieved and Maintained a Testosterone Castration (Testosterone Level of <50 [Nanograms per Deciliter] ng/dL and <20 ng/dL) | Cohorts 1, 2, and 3: Days 29 to 85
Number of Participants who Maintained a Testosterone Castration (Testosterone Level of <50 ng/dL and <20 ng/dL) | Cohort 3: Days 29 to 169
Time to Achieve Testosterone Castration (Testosterone Level of <50 ng/dL and <20 ng/dL) | Cohorts 1 and 2: Day 1 up to Day 85; Cohort 3: Day 1 up to Day 169
Number of Participants who Experience Local Reactions Categorized as Erythema, Swelling, and Induration at the Injection Site | Cohorts 1 and 2: Immediately, at 2 and 24 hours post-injection on Day 1; Cohort 3: Immediately, at 2 and 24 hours post-injection on Days 1 and 85
Number of Participants who Experience Pain at Injection Site | Cohorts 1 and 2: Immediately, at 2 and 24 hours post-injection on Day 1; Cohort 3: Immediately, at 2 and 24 hours post-injection on Days 1 and 85
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) By Severity | Cohorts 1 and 2: Up to Day 169; Cohort 3: Up to Day 197
Number of Participants With Related TEAEs, Serious TEAEs, Adverse Events of Special Interest (AESIs), TEAEs Leading to Treatment Delay, and/or Discontinuation, and Death | Cohorts 1 and 2: Up to Day 169; Cohort 3: Up to Day 197
Number of Participants With Clinically Significant Abnormalities in Laboratory, Vital Signs, and Electrocardiogram (ECG) Parameters | Cohorts 1 and 2: Up to Day 169; Cohort 3: Up to Day 197
Percent Change From Baseline in Serum Prostate-Specific Antigen (PSA) Over Time | Cohorts 1 and 2: Baseline up to Day 85; Cohort 3: Baseline up to Day 169
Change From Baseline of Serum Luteinizing Hormone (LH) Over Time | Cohorts 1 and 2: Baseline up to Day 85; Cohort 3: Baseline up to Day 169
Change From Baseline in Serum Follicle-Stimulating Hormone (FSH) Over Time | Cohorts 1 and 2: Baseline up to Day 85; Cohort 3: Baseline up to Day 169

CONTACTS AND LOCATIONS:
Locations (37):
- United States (23):
  - Urologic Surgeons of Arizona, Mesa, Arizona
  - East Valley Urology Center of Arizona, Queen Creek, Arizona
  - Bakersfield Institute of Advanced Urology, Bakersfield, California
  - Grimaldi Urology, Chula Vista, California
  - Valley Urology, Fresno, California
  - Urology Group of Southern California, Los Angeles, California
  - Advanced Urology, Los Angeles, California
  - Tower Urology,, Los Angeles, California
  - Alarcon Urology Center, Montebello, California
  - Urology Center of Southern California, Murrieta, California
  - Pasadena Urological Medical Group, Pasadena, California
  - AP Medical Research, Miami, Florida
  - Biogenix Molecular, Miami, Florida
  - First Urology- Jeffersonville, Jeffersonville, Indiana
  - GU Research Network/Wichita Urology Group, Wichita, Kansas
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - New York Cancer and Blood Specialists, Shirley, New York
  - Associated Urologists of North Carolina, Raleigh, North Carolina
  - Oregon Urology Institut, Springfield, Oregon
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology Clinics of North Texas, Dallas, Texas
  - Urology of Virginia, Virginia Beach, Virginia
  - Summit Cancer Centers of North Spokane, Spokane, Washington
- Belgium (3):
  - University Hospital Gent, Ghent
  - AZ Groeninge, Kortrijk
  - AZ Delta, Roeselare
- France (6):
  - CHU Angers, Angers
  - CHRU de Brest - Hopital Morvan, Brest
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges Francois Leclerc, Dijon
  - CHU de Nantes - Hôtel Dieu, Nantes
  - AP-HP Hopital Pitie-Salpetriere, Paris
- Spain (5):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Clinico San Carlos, Madroñera
  - Corporacio Sanitaria Parc Tauli - Hospital de Sabadell, Sabadell
  - Instituto Valenciano de Oncologia, Valencia

IPD SHARING:
Plan to Share IPD: No